CLINICAL TRIAL: NCT02762370
Title: A Double-Blind, Randomized, Parallel Group Comparison of the Effects of FX006 and TCA IR (Triamcinolone Acetonide Suspension) on Blood Glucose in Patients With Osteoarthritis of the Knee and Type 2 Diabetes Mellitus
Brief Title: Study to Assess the Effects of FX006 on Blood Glucose in Patients With OA of the Knee and Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2015-010
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee; Type 2 Diabetes Mellitus
Keywords: osteoarthritis; knee; pain; diabetes; intra-articular; injection; corticosteroid
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus, Type 2; Osteoarthritis; Pain; Diabetes Mellitus | interventions — FX006; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FX006 32 mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release Formulation
  Interventions: Drug: FX006 32 mg
- TCA IR 40 mg (Active Comparator): Single 1 mL intra-articular (IA) injection Immediate-release Formulation
  Interventions: Drug: TCA IR 40 mg

INTERVENTIONS:
Drug: FX006 32 mg — Single 5 mL IA injection
  Other Names: Zilretta
  Arms: FX006 32 mg
Drug: TCA IR 40 mg — Single 1 mL IA injection
  Other Names: Kenalog®-40 Injection; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
The purpose of this study was to compare the effects of FX006 and Triamcinolone Acetonide Injectable Suspension, United States Pharmacopeia (USP) (referred to as TCA IR in the protocol) on blood glucose (BG) in patients with osteoarthritis (OA) of the knee and Type 2 diabetes mellitus (DM).

DETAILED DESCRIPTION:
This study employed a double-blind, randomized, parallel group, single dose design to explore the pharmacodynamic effects on BG levels in type 2 diabetics following IA administration of 32 mg FX006 compared to 40 mg TCA IR. The study was conducted in male and female patients ≥40 years of age with OA of the knee and type 2 DM not managed by injectable agents. In order to be eligible for study participation, patients were to be treated with 1 or 2 oral agents and have hemoglobin A1c (HbA1c) levels between 6.5%-9.0%.

Approximately 36 patients were planned to be randomized and treated to ensure there were at least 30 evaluable patients (15 patients on FX006 and 15 patients on TCA IR). Patients were randomized to 1 of 2 treatment groups (1:1) and treated with a single IA injection of either:

* 32 mg FX006 (18 patients) or
* 40 mg TCA IR (18 patients)

BG levels in each patient were evaluated for a total of 3 weeks (1 week prior to IA injection and 2 weeks post IA injection). After a screening visit, patients' BG levels were measured using a Dexcom Z4 Platinum Professional™ continuous glucose monitor (CGM) device, set to blinded mode, for up to 1 week pre-injection and for 2 weeks post injection using the same blinded CGM device. Patients also were provided with a Bayer Contour™ standard glucose measuring meter in order to perform the necessary calibrations per the manufacturer's recommendations. A final safety visit was planned at 6 weeks post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female ≥40 years of age
* Type 2 diabetes mellitus for at least 1 year prior to Screening and not managed with injectable agents (e.g. insulin or insulin analogs, exenatide, pramlintide, liraglutide)
* Currently treated with 1 or 2 oral agents for diabetes, with stable doses for at least 2 months
* HbA1c ≥6.5% and ≤ 9.0%
* Currently meets American College of Rheumatology (ACR) Criteria (clinical or radiological) for OA.
* Symptoms associated with OA of the knee for ≥ 6 months prior to Screening
* Index knee pain on most days (>15) over the last month (as reported by the patient)
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of protocol-specified restricted medications during the study
* Willingness to wear a CGM device uninterrupted for 24 hours per day throughout the study, remain with receiving range and comply with calibration requirements
* Accustomed to using a Standard Blood Glucose Measuring device by finger stick

Exclusion Criteria:

* Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis or arthritis associated with inflammatory bowel disease
* History of infection in the index knee joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee within 1 month of Screening
* Presence of surgical hardware or other foreign body in the index knee
* Unstable joint (such as a torn anterior cruciate ligament) within 12 months of screening
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* IV or intramuscular (IM) corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Any other IA investigational drug/biologic within 6 months of Screening
* Prior use of FX006
* Use of acetaminophen, or acetaminophen containing products
* Current use of a continuous glucose monitoring device
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (8):
- United States (8):
  - Anaheim, California
  - El Cajon, California
  - North Hollywood, California
  - Duncansville, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Russell SJ, Sala R, Conaghan PG, Habib G, Vo Q, Manning R, Kivitz A, Davis Y, Lufkin J, Johnson JR, Kelley S, Bodick N. Triamcinolone acetonide extended-release in patients with osteoarthritis and type 2 diabetes: a randomized, phase 2 study. Rheumatology (Oxford). 2018 Dec 1;57(12):2235-2241. doi: 10.1093/rheumatology/key265. PMID 30203101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for study eligibility at 9 study centers in the United States (US).
Pre-assignment Details: Patients were Randomized within 21 days of Screening.
Groups:
- FX006 32 mg: 18 subjects received FX006 32 mg as a single 5 mL intra-articular (IA) injection
- TCA IR 40 mg: 15 subjects received triamcinolone acetonide injectable suspension, immediate release (TCA IR) 40 mg as a single 1 mL IA injection
Period: Overall Study
Arm/Group | FX006 32 mg | TCA IR 40 mg
Started | 18 | 15
Completed | 17 | 15
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- FX006 32 mg: FX006: Single 5 mL IA injection
- TCA IR 40 mg: TCA IR: Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 32 mg | TCA IR 40 mg | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (5.76) | 60.3 (10.38) | 61.2 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Average Blood Glucose (mg/dL)
Description: Average blood glucose was analyzed with a mixed model for repeated measures (MMRM)
Time Frame: Baseline and 72 Hours post intra-articular (IA) injection
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- FX006 32 mg: Drug: FX006 Single intra-articular injection
  FX006 32 mg
- TCA IR 40 mg: Drug: TCA IR Single intra-articular injection
  TCA IR 40 mg
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
mg/dL | 14.66 (7.032) | 33.88 (6.612)
Statistical Analysis 1: Comparison: FX006 32 mg vs TCA IR 40 mg; Test type: Superiority; p = 0.0452, t-test, 2 sided

2. Secondary Outcome: Percent Time Blood Glucose Less Than 70 mg/dl, 70 - 180 mg/dl, 180.1 - 250.0 mg/dl, 250.1 - 350.0 mg/dl, and Greater Than 350.0 mg/dl
Description: The glycemic variability was calculated as the coefficient of variation (CV) of the hourly averages in each of these time periods: Hour 1-24, Hour 1-48, Hour 1-72, Hour 1-168, and Hour 1-360. The % CV for each patient was derived using the formula: (SD/mean)*100, using the values for each hourly average glucose measurement over the time period. Average % CV in the FX006 40 mg group was compared to the TCA IR 40 mg group using a linear model (ANCOVA) with fixed effects for treatment group. Model covariates were study center and baseline (72-hour) blood glucose average.
Time Frame: Baseline to Days 1-3
Measure: Number; unit: Percentage of time
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
Percentage of time
  Less than 70 | 2.2 | 0.4
  70 - 180 | 63.3 | 49.7
  180.1 - 250.0 | 23.7 | 24.5
  250.1 - 350.0 | 9.5 | 21.1
  Greater than 350.0 | 1.3 | 4.3

3. Secondary Outcome: Glycemic Variability Coeffecient of Variation (CV)
Description: as for outcome 2
Time Frame: Baseline to 72 hours post injection (hourly average blood glucose measurement over the time period)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
mg/dL | 22.43 (1.434) | 27.05 (1.349)

4. Secondary Outcome: Area Under the Effect (AUE) Curves for Average Blood Glucose - FX006 Versus TCA IR
Time Frame: Baseline to 72 hours post injection (-72 hr, 0 hr, and 1, 2, 3, 7, and 15 days post-dose)
Measure: Least Squares Mean (Standard Error); unit: hr*mg/dL
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
hr*mg/dL
  Baseline (Hour -72 to Hour -1) | 22089.0 (775.19) | 23669.1 (728.86)
  Day 1 | 3703.3 (239.62) | 4483.2 (225.30)
  Days 1-2 | 7902.6 (442.21) | 9251.7 (415.78)
  Days 1-3 | 11772.3 (652.17) | 12950.9 (613.20)
  Days 1-7 | 27245.7 (1615.93) | 25987.0 (1519.37)
  Days 1-15 | 52112.8 (2966.97) | 49532.2 (2789.67)

5. Other Pre Specified Outcome: Percent Time Blood Glucose Less Than 70 mg/dl, 70 - 180 mg/dl, 180.1 - 250.0 mg/dl, 250.1 - 350.0 mg/dl, and Greater Than 350.0 mg/dl
Time Frame: Baseline to Days 1-2
Measure: Number; unit: Percentage of time
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
Percentage of time
  Less than 70.0 | 1.2 | 0.3
  70.0 - 180.0 | 64.1 | 42.7
  180.1 - 250.0 | 23.0 | 27.4
  250.1 - 350.0 | 9.9 | 25.2
  Greater than 350.0 | 1.7 | 4.4

6. Other Pre Specified Outcome: Change From Baseline for Maximum Blood Glucose: Baseline Average Blood Glucose (Hour -72 to Hour -1) to Maximum Blood Glucose (Hour 1 to Hour 72) for FX006 32 mg Relative to TCA IR 40 mg
Time Frame: Baseline (Hour -72 to Hour -1) to Hour 1 to Hour 72
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
mg/dL | 110.04 (10.084) | 158.46 (9.481)

7. Other Pre Specified Outcome: Change in Average Blood Glucose From Baseline (Hour -48 to Hour -1) to Hour 1 to Hour 48 for FX006 32 mg Relative to TCA IR 40 mg.
Time Frame: Baseline (Hour -48 to Hour -1) to Hour 1 to Hour 48
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 18 | 15
mg/dL | 16.33 (8.791) | 43.62 (8.255)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 1 (following IA administration) through Day 43.
Arm/Group | FX006 32 mg | TCA IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 2/18 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=18) | TCA IR 40 mg (N=15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Subsequent to completion of clinical studies extensive testing was performed to assess the actual FX006 dose delivered. It was determined that the FX006 delivered dose to the patient from an FX006 40 mg vial is 32 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes